CLINICAL TRIAL: NCT04329026
Title: The Usefulness of Smart-glasses During the Ultrasound-guided Radial Arterial Catheterization in Pediatric Patients: a Randomized Controlled Trial
Brief Title: Smart-glasses During the US-guided Radial Arterial Catheterization in Pediatric Patients: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Smart Glass A-line
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Arterial Line
Keywords: Radial Artery; Vascular Catheters; Smart Glassess
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Glasses (Experimental): The real-time ultrasound image is displayed through head-mounted display Moverio BT-300 (Epson Inc., USA) during the radial arterial cannulation.
  Interventions: Device: Smart glasses
- Control (Placebo Comparator): The real-time ultrasound image is displayed by the ultrasound machine's monitor during the radial arterial cannulation.
  Interventions: Device: Control

INTERVENTIONS:
Device: Smart glasses — The real-time ultrasound image is displayed through head-mounted display Moverio BT-300 (Epson Inc., USA) during the radial arterial cannulation.
  Arms: Smart Glasses
Device: Control — The real-time ultrasound image is displayed by the ultrasound machine's monitor during the radial arterial cannulation.
  Arms: Control

SUMMARY:
The primary objective of the study is to evaluate the effect of smart glasses (Head-mounted display Moverio BT-300 (Epson Inc., USA)) on the first-attempt success rate of radial artery cannulation in pediatric patients. This study hypothesizes that the use of smart glasses improves the hand-eye coordination and the first-attempt success rate of radial artery cannulation. This is a single-center, randomized, placebo-controlled study comparing the real-time ultrasound image through smart glasses (intervention group) or the ultrasound machine's monitor (control group) during the radial arterial cannulation in pediatric patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Arterial cannulation for hemodynamic monitoring, multiple blood sample

Exclusion Criteria:

* Unstable vital sign, significant arrhythmia or hypotension, Shock
* High risk of peripheral ischemia
* Skin disease, infection, hematoma, recent cannulation at radial artery

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | During radial artery cannulation (up to 1 hour)
  Success at the first skin puncture

SECONDARY OUTCOMES:
Size of radial artery | Before and after subcutaneous injection of drugs (up to 1 hour)
  Internal diameter of radial artery
depth of radial artery | During radial artery cannulation (up to 1 hour)
  depth of radial artery from the skin
Overall attempt | During radial artery cannulation (up to 1 hour)
  Number of attempt of radial artery cannulation
Overall Procedure time | During radial artery cannulation (up to 1 hour)
  From needle puncture, to Arterial waveform
Overall success rate | During radial artery cannulation (up to 1 hour)
  Success within 2 skin puncture and within 10 minutes at the chosen radial artery
Malfunction of radial artery catheter | After radial artery cannulation assessed during anesthesia (up to 24 hour)
  Malfunction of Invasive blood pressure monitoring, Sampling
Complication rate | After radial artery cannulation assessed up to PACU, PICU stay (up to 24 hour)
  Hematoma, Distal ischemia, Spasm accessed by ultrasound
Operator's satisfaction | During radial artery cannulation (up to 1 hour)
  Operator's satisfaction, 5 scale (Worst, Poor, Acceptable, Good, Best)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White L, Halpin A, Turner M, Wallace L. Ultrasound-guided radial artery cannulation in adult and paediatric populations: a systematic review and meta-analysis. Br J Anaesth. 2016 May;116(5):610-7. doi: 10.1093/bja/aew097. PMID 27106964
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Lee WJ, Kim HS. Posterior Tibial Artery as an Alternative to the Radial Artery for Arterial Cannulation Site in Small Children: A Randomized Controlled Study. Anesthesiology. 2017 Sep;127(3):423-431. doi: 10.1097/ALN.0000000000001774. PMID 28682811
- [Background] Cuper NJ, de Graaff JC, Hartman BJ, Verdaasdonk RM, Kalkman CJ. Difficult arterial cannulation in children: is a near-infrared vascular imaging system the answer? Br J Anaesth. 2012 Sep;109(3):420-6. doi: 10.1093/bja/aes193. Epub 2012 Jun 26. PMID 22735300
- [Background] Ishii S, Shime N, Shibasaki M, Sawa T. Ultrasound-guided radial artery catheterization in infants and small children. Pediatr Crit Care Med. 2013 Jun;14(5):471-3. doi: 10.1097/PCC.0b013e31828a8657. PMID 23628835
- [Background] Song IK, Choi JY, Lee JH, Kim EH, Kim HJ, Kim HS, Kim JT. Short-axis/out-of-plane or long-axis/in-plane ultrasound-guided arterial cannulation in children: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):522-7. doi: 10.1097/EJA.0000000000000453. PMID 26986774
- [Background] Maruyama K, Watanabe E, Kin T, Saito K, Kumakiri A, Noguchi A, Nagane M, Shiokawa Y. Smart Glasses for Neurosurgical Navigation by Augmented Reality. Oper Neurosurg. 2018 Nov 1;15(5):551-556. doi: 10.1093/ons/opx279. PMID 29373710